CLINICAL TRIAL: NCT07259759
Title: JURA Study - Observational First-in-human Feasibility Study
Acronym: JURA
Status: Recruiting | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1145917C
Record Dates: First submitted 2025-09-25; First posted 2025-12-02 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Imaging
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JURA Group: Visualization of organs, structures and tissue of interest using the JURA System during a surgical procedure. The surgical procedure itself will be conducted exclusively following the site standard of care.
  Interventions: Device: Visualization / Imaging

INTERVENTIONS:
Device: Visualization / Imaging — Visualization / Imaging of organs, structures and tissue of interest using the JURA system such as for example spleen, anastomosis of colon, omental fat, pancreas

SUMMARY:
Evaluate the functionality of the JURA System v. 1.0

DETAILED DESCRIPTION:
Evaluate the functionality of the JURA System v. 1.0 in humans under real clinical conditions in the operating room

ELIGIBILITY:
Key Inclusion Criteria:

1. Men and women ≥ 18 years of age
2. Patient scheduled for an elective abdominal minimal invasive surgery

Key Exclusion Criteria:

1. Pregnancy, or positive pregnancy test for women prior to menopause or breastfeeding women
2. Individuals who are unable to fully understand all aspects of the study as relevant to the decision to participate (mentally or verbally), or who could be manipulated or unduly influenced due to of a compromised position, expectation or benefits or fear or retaliation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women above the age of 18 year, scheduled for an elective abdominal minimal invasive surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Image quality of the JURA System v. 1.0 in humans | Intra-Operative
  Image quality of the JURA System v. 1.0 in humans using an image quality assessment score

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, ZA, Netherlands

IPD SHARING:
Plan to Share IPD: No